CLINICAL TRIAL: NCT06503510
Title: The Role of the Interleukin-13 Pathways on Pain and Itch Sensitivity in Patients With Atopic Dermatitis and Healthy Volunteers
Brief Title: Role of Interleukin-13 Pathways on Pain and Itch Sensitivity
Acronym: IL-13
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Silvia Lo Vecchio, Professor, Aalborg University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N-20240029
Record Dates: First submitted 2024-07-10; First posted 2024-07-16 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-01

CONDITIONS: Itch
MeSH Terms: conditions — Pruritus | interventions — Histamine; bovine adrenal medulla 8-22

STUDY DESIGN:
Intervention Model Description: Each participant will be treated with Lebrikizumab and will receive 3 pruritogens: Histamine, cowhage and BAM8-22.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Lebrikizumab (Experimental): The initial doses will be subcutaneous Lebrikizumab 500 mg (two 250 mg injections) at both week 0 (baseline) and week 2, followed by 250 mg administered subcutaneously at week 4.
  Interventions: Other: Histamine; Other: Cowhage; Other: bovine adrenal medulla (BAM8-22)

INTERVENTIONS:
Other: Histamine — A small drop of histamine dihydrochloride (1%, in saline) will be applied to a previously determined area on the volar forearm followed by a prick through the drop.
Other: Cowhage — Approximately 30-35 cowhage spicules will be manually inserted into the subject's skin.
Other: bovine adrenal medulla (BAM8-22) — A small drop of BAM8-22 solution will be applied to a previously determined area on the volar forearm followed by a prick through the drop.

SUMMARY:
Atopic dermatitis (AD) is as chronic, inflammatory skin disorder affecting 20% of the world's population. Intense itch and skin pain are the main symptoms. Research has shown that the proteins interleukins are involved in inflammation and itch in atopic dermatitis. The medicinal product called Lebrikizumab, used for treatment of AD, has shown to block the interleukin called IL-13. The purpose of this experiment is to evaluate the role of IL-13 in itch in both healthy subjects and people with atopic dermatitis.

DETAILED DESCRIPTION:
Atopic dermatitis (AD) is as chronic, inflammatory skin disorder affecting 20% of the world's population. Intense itch and skin pain are the main symptoms. Research has shown that the interleukin-13 is involved in inflammation and itch in atopic dermatitis by increasing the neuronal sensitivity to pruritogens. However, the physiological mechanisms by which IL-13 increases the itch sensitivity are unclear. The aim of this project is to use, for the first time in humans, the monoclonal antibody Lebrikizumab that inhibits IL-13 with high affinity as a novel experimental tool to modulate the IL-13 pathway and evaluate its role in the transmission and processing of itch and pain.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* 18-60 years

Exclusion Criteria:

* Pregnancy or lactation
* Drug addiction defined as any use of cannabis, opioids, or other drugs
* Previous or current history of neurological, dermatological (e.g., AD, psoriasis, etc.), immunological, musculoskeletal, cardiac disorder, or psychiatric diagnoses that may affect the results (e.g., neuropathy, muscular pain in the upper extremities, anxiety, depression, schizophrenia, etc.)
* Moles, wounds, scars, or tattoos in the area to be treated or tested
* Current use of medications that may affect the trial such as antihistamines and pain killers (use of antihistamines should be discontinued 72 hours before the experiment and all topical agents and emollients should be discontinued 24 hours before the experiment).
* Use of systemic and topical corticosteroids
* Consumption of alcohol or painkillers 24 hours before the study days and between these
* Acute or chronic pain
* Participation in other trials within one week of study entry (four weeks in the case of pharmaceutical trials)
* Lack of ability to cooperate

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Measuring itch by computerized Visual Analog Scale Scoring | 1 minute after every itch induction
  The subjects will be asked to rate the sensation of itch on a 100 mm VAS scale ranging from 0 to 100 where 0 indicates "no itch" and 100 indicates "worst itch imaginable".
Measuring pain by computerized Visual Analog Scale Scoring | 1 minute after every itch induction
  The subjects will be asked to rate the sensation of pain on a 100 mm VAS scale ranging from 0 to 100 where 0 indicates "no pain" and 100 indicates "worst pain imaginable".
Superficial blood perfusion | Baseline
  Superficial blood perfusion (SBP) is measured by a Speckle contrast imager
Superficial blood perfusion | 10 minute after every itch induction
  Superficial blood perfusion (SBP) is measured by a Speckle contrast imager
Wheal reaction | 10 minute after every itch induction
  Wheal reaction measurement will be conducted immediately after the removal of pruritogens by measuring the longest diameter with a ruler.
Average pruritis and pain numerical rating scale (NRS) | Baseline
  The subject will be asked to retrospectively rate the average and worst itch/pain on an 11-point scale ranging from 0 to 10 (0 = no pain and 10 = worst imaginable pain)experience they had during the last 7 days.
Skin peak pain numerical rating scale (SPP-NRS) | Baseline
  According to the SPP-NRS, the subject will be asked about "worst skin pain" they felt in the past 24 hours on an 11-point scale ranging from 0 to 10 (0 = no pain and 10 = worst imaginable pain)
Peak pruritus numerical rating scale (PP-NRS) | Baseline
  The subject will be asked about the "worst itch" they felt in the past 24 hours on an 11-point scale ranging from 0 to 10 (0 = no itch and 10 = worst imaginable itch)
Mechanically evoked itch (MEI) | Baseline
  MEI is measured by using mildly pruritic, non-painful von Frey nylon filaments of a predetermined intensity (generally 5-30 miliNewton of force).
Mechanically evoked itch (MEI) | 10 minutes after every itch induction
  MEI is measured by using mildly pruritic, non-painful von Frey nylon filaments of a predetermined intensity (generally 5-30 miliNewton of force).

SECONDARY OUTCOMES:
Mechanical Pain Thresholds (MPT) | Baseline
  This test is conducted using a pinprick set. The set consists of 7 needles each with a diameter of 0.6 mm and different force applications: 8, 16, 32, 64, 128, 256, and 512 mN.
Mechanical Pain Sensitivity (MPS) | Baseline
  This test is conducted with the same pinprick set used to test the MPT.
Pressure Pain Thresholds (PPT) | Baseline
  Pressure will be applied by a handheld electronic pressure algometer (Somedic AB, Stockholm, Sweden) on to the supinator muscle on the left forearm.
Cold Detection Thresholds (CDT) | Baseliene
  The tests of thermal sensation will all be conducted using a TSA2 (Medoc Ltd, Israel) thermal sensory testing device
Warm Detection Thresholds (WDT) | Baseline
  The tests of thermal sensation will all be conducted using a TSA2 (Medoc Ltd, Israel) thermal sensory testingdevice
Cold Pain Thresholds (CPT) | Baseline
  The tests of thermal sensation will all be conducted using a TSA2 (Medoc Ltd, Israel) thermal sensory testing device
Heat Pain Thresholds (HPT) | Baseline
  The tests of thermal sensation will all be conducted using a TSA2 (Medoc Ltd, Israel) thermal sensory testing device
Pain to Supra-threshold Heat Stimuli (STHS) | Baseline
  The tests of thermal sensation will all be conducted using a TSA2 (Medoc Ltd, Israel) thermal sensory testing device

CONTACTS AND LOCATIONS:
Locations (3):
- Denmark (3):
  - Aalborg University, Gistrup, Aalborg
  - CNAP, Gistrup, Aalborg
  - Aalborg University, Aalborg, Denmark